# Official Title of the study: Evaluation of the Efficacy of Polybutester Suture on Postoperative Complications in Lower

Date: 11, Feb 2022

# 1. Corresponding author: Levent Cigerim

Address: Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and

Maxillofacial Surgery, Van, Turkey Postal Code: 65080

Phone: +905321633287 Office Phone: 904322251744 Fax: +904322251747.

Email: levent139@hotmail.com

# 2. Zeynep Dilan Orhan

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery

Email: zeynepdilanorhan@gmail.com,

Phone: +905425525525

#### CONSENT FORM FOR RESEARCH

### Dear patient,

Please read this document carefully and listen carefully to what we have said. Detailed information about the research; Detailed information about your rights, benefits and risks of the research can be found in this document. The purpose of these statements is to inform you about your health. Please indicate what you do not understand, your questions will be explained in detail. You can leave the research at any stage of the research if you think that your questions are not adequately explained after you accept to participate in the research or for any other reason. During the research period, the health problems arising from our research will be treated in our hospital immediately. You will not be charged an additional fee for participating in this research, nor will you be paid. Thank you for participating in our research.

## Name of the Study:

The subject, purpose, method, time and process to be used of the research: Our research is about the effect of suture to be used in impacted wisdom tooth extraction on postoperative complaints. Patients coming for impacted tooth extraction will be divided into two groups and the effectiveness of the polybutester and polypropylene suture to be used on postoperative complaints will be evaluated. In the evaluation of this activity, you will be given a form for pain and you will be asked to fill in this form. Evaluation of other effects will be done by measuring methods in our clinic.

**Suggested procedure/process for research:** In our research, the recommended procedure/process for each operation is 1 week. Evaluations in our clinic will be made before the operation, 2 days after the operation and 7 days after the operation.

Damages or possible risks that may occur during the research: (Complications/complaints that may occur here can be seen in routine impacted wisdom teeth surgeries.) Pain, swelling and/or redness, discomfort in the surgical area, limitation in mouth opening, bleeding (during/after the procedure), infection, redness and cracking due to stretching in the corners of the mouth, Temporary or permanent loss of sensation in the lip and/or tongue, soft tissue injuries, damage to adjacent teeth and surrounding tissues, protrusion/breakage of the jaw, entry of teeth or foreign objects into the respiratory tract, trauma to the temporomandibular joint, side effects due to drugs (allergy, nausea, vomiting), diarrhea, gastrointestinal system problems, dizziness, anxiety, numbness, fatigue)

Study-specific risks during the study: None.

Possible benefits of the research: Complaints experienced by patients after impacted tooth

extraction will be reduced.

**Anesthesia:** Local anesthesia is used to control pain during the treatment.

**Funding of the research:** You will not be charged an additional fee for participating in this research and you will not be paid any money.

Evaluation of the Efficacy of Polybutester Suture on Postoperative

| Complications in Lower Impacted Third Molar Surgery |
|---|
| Dear patient/ participant/, please read the following articles |
| carefully and fill in the relevant blank or tick the relevant box |
| 1. I was invited to the research after I received the preliminary information about the research explained in a clear and simple way and after reading the consent form in my hand. subject invitation; I agreed. I did not accept. 2. I have read and listened to the points to be considered in the research. I asked my questions |
| 3. Provided that my identity is kept confidential and used only for educational and research purposes, I may be photographed during the intervention/treatment to be applied to me, that my data can be used retrospectively or recorded. I allow I do not allow. 4. I learned the benefits and possible risks of diagnostic interventions, medical and surgical treatments, and the procedures to be done. I agree. I do not accept. |
| 5. Since I can't read/write the research information process or I don't want to decide on my own |
| joined |
| 6. The data received by me regarding the research will be kept confidential, i know know 7. I have the right to withdraw from the research at any time, (I know, I don't know) 8. I will not charge/pay any fee as a result of the research. (I know, I don't know) 9. If a medical risk arises, free medical treatment will be provided. (I know, I don't know) 10. The possible benefits of the research result in detail. (I know, I don't know) 12. When I encounter a health problem during the research; at any hour, (I know that I can call Dt. Zeynep Dilan Orhan at 0432 225 17 44 (work) / 0536 699 85 27 (mobile) at YYU Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery. |
| The Participant's and/or Legal Representative to Get Consent in Emergency Situations |
| Date: Name surname: Date of birth: |
| Address: |
| Signature : |

# Name-Surname of the Physician Responsible for the Research:

Associate Professor Levent Cigerim

**Institution Registration Number: 5086** 

Signature :